CLINICAL TRIAL: NCT06692387
Title: STEPWISE Parkinson: A Smartphone Based, Titrated Exercise Solution for Patients With Parkinson's Disease in Daily Life - Pilot Study
Brief Title: A Smartphone Based, Titrated Exercise Solution for Patients With Parkinson's Disease in Daily Life: Pilot Study
Acronym: STEPWISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL74352.091.20
Record Dates: First submitted 2020-07-03; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Movement Disorders; Parkinson Disease
Keywords: Physical activity; Walking; Exercise; Parkinson Disease; Locomotion; Motivational application
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active control group (Active Comparator): Ten people will be encouraged to increase their physical activity level, measured in step counts on the patients' own smartphone, with 10% compared to their own baseline level.
  Interventions: Behavioral: Step count increase with the use of a motivational application
- Step count increase 50% (Experimental): Ten people will be encouraged to increase their physical activity level, measured in step counts on the patients' own smartphone, with 50% compared to their own baseline level.
  Interventions: Behavioral: Step count increase with the use of a motivational application
- Step count increase 100% (Experimental): Ten people will be encouraged to increase their physical activity level, measured in step counts on the patients' own smartphone, with 100% compared to their own baseline level.
  Interventions: Behavioral: Step count increase with the use of a motivational application

INTERVENTIONS:
Behavioral: Step count increase with the use of a motivational application — The motivational app will encourage people to increase their physical activity for a short period of time (one month). Different treatment arms will receive different physical activity goals. People will get feedback and be motivated based on their own baseline level and actual activity level.

SUMMARY:
The aim of this pilot randomized controlled trial is to test whether it's feasible to increase participants' step counts within four weeks with a developed motivational smartphone application. If this is feasible, then we can proceed to test the app in a large, long-term randomized clinical trial.

DETAILED DESCRIPTION:
Rationale: Exercise affords health benefits for people with Parkinson's disease (PD), but implementing exercise in daily life remains challenging. Moreover, many training programs are not very scalable. The investigators take an important step forward by developing and studying an innovative and fully decentralized smartphone-based program to increase long-term physical activity in people with PD in daily life.

Objective: The aim of this pilot study is to investigate whether the developed smartphone app can increase physical activity in people with PD for a short period of time (one month). The secondary aim is to study the usability and enjoyment of the app and the potential effects of an increase in physical activity on physical fitness, motor- and non-motor functioning.

Study design: Pilot double-blind randomized controlled intervention study.

Study population: A total of 30 Dutch people with PD who have no other medical conditions that markedly hamper mobility, no cognitive impairments that make it difficult to use a game on the smartphone and possess a suitable smartphone, will be recruited.

Intervention: Participants will be randomized into one of three groups. All groups will be encouraged to increase their physical activity level, measured in step counts on the participants' own smartphone, with a different percentage: (a) an increase in step count of 10% (active control group, N = 10), (b) in increase in step count of 50% (experimental group 1, N = 10), or (c) an increase in step count of 100% (experimental group 2, N = 10), compared to their baseline level.

ELIGIBILITY:
Inclusion Criteria:

1. idiopathic PD
2. Hoehn and Yahr 1-3
3. able to understand the Dutch language
4. able to walk independently
5. less than 30 minutes of sports/outdoor activities per day (LASA Physical Activity Questionnaire, LAPAQ)
6. less than 7,000 steps/day during 1-week baseline

Exclusion Criteria:

1. weekly falls in the previous 3 months
2. medical conditions that hamper mobility
3. living in a nursing home
4. cognitive impairments that hamper use of the motivational app on the smartphone (Montreal Cognitive Assessment, MoCA <26)
5. not in the possession of a suitable smartphone (Iphone 5S or newer with iOS 10 or higher or Android 4.1 or newer)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the last week of the intervention in step count | Change from baseline to the last week of the intervention (week 4)
  Step counts measured continuously with patients' own smartphone

SECONDARY OUTCOMES:
Change in PD motor symptoms | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) part 3. Range: 0-132. Higher scores indicate worse function.
Change in Motor functioning in daily life | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) part 2. Range: 0-52. Higher scores indicate worse function.
Change in Physical fitness | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Meters walked during the six minute walk test (6MWT). Higher scores indicate better function.
Change in Mobility | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Timed Up and Go Test, number of seconds to complete standing up from a chair, walk 3 meters, turn, walk 3 meters back and sit down. Higher scores indicate worse function.
Change in Balance | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  The mini balance evaluation system (mini-BEST) is a 14-item, 3 points ordinal rating scale (0-2 points) to evaluate balance performance in 4 subcategories: anticipatory postural control, reactive postural control, sensory orientation and stability in gait. The attainable scores ranges from 0-28 points, in which a higher score indicates better balance.
Change in Gait speed | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  The ten meter walk test (10MWT) is a standardised and recommended measurement of walking velocity. The number of seconds it takes to walk ten meters is recorded. Higher scores means worse function.
Change in Fear of falling | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Falls Efficacy Scale International [FES-I]. Range: 16-64. Higher score reflects higher fear of falling
Change in Handgrip strength | Change from baseline to post-intervention in the first week after week 4 (week 5)
  Handgrip strength measured with a dynamometer. Higher scores mean better function.
Change from baseline to post-intervention after week 4 in Self-reported physical activity level | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  LASA Physical Activity Questionnaire (LAPAQ). Range: 0-no maximum. Higher score reflecting more time spent in physical activities;
Change from baseline to post-intervention after week 4 in Global PD non-motor symptoms | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) part 1. Range: 0-52. Higher scores mean worse function.
Change in Cognition | Change from baseline to post-intervention in the first week after week 4 (week 5)
  Montreal Cognitive Assessment (MoCA). Range: 0-30. Higher scores reflect better cognition.
Change in Depression and anxiety | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Hamilton Anxiety and Depression Scale; HADS; Minimum score = 0 (no anxiety or depression), maximum score = 42 (most anxiety or depression). Higher scores mean more anxiety/depression.
Change in Apathy | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Abbreviated version of the Apathy Evaluaton Scale; AES-12PD. Range 12-48. Higher scores indicate better function.
Change in Sleep | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Scales for Outcomes in Parkinson's Disease-Sleep; SCOPA-SLEEP. Range: 0-33. Higher scores reflect worse sleep.
Change in Autonomic dysfunction | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Scales for Outcomes in Parkinson's Disease-Autonomic questionnaire; SCOPA-AUT. Range: 0-69. Higher scores indicate more problems with autonomic function.
Change in Health-related quality of life | Change from baseline to the post-intervention visit in the first week after week 4 (week 5)
  Parkinson's Disease Questionnaire; PDQ-39. Range: 0-100. Lower scores reflecting a better health-related quality of life

OTHER OUTCOMES:
System Usability (SUS) | After the post-intervention visit in the first week after week 4 (week 5)
  Usability of the STEPWISE application as assessed by the Dutch version of the System Usability Scale (SUS) at 5 weeks (follow-up). Range 0-100. Higher scores indicate better usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands